CLINICAL TRIAL: NCT02387632
Title: Airway Pressure During Humidified High Flow Nasal Cannula Therapy in Children
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Karen Choong, Associate Professor, McMaster University
Other Study IDs: 15-079
Record Dates: First submitted 2015-03-08; First posted 2015-03-13 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2015-11

CONDITIONS: Bronchiolitis; Pneumonia; Bronchial Asthma
MeSH Terms: conditions — Bronchiolitis; Pneumonia; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Humidified High Flow Nasal Cannula (HHFNC) is a new modality of respiratory support for children with respiratory failure. Despite its extensive use in pediatric and adult population, the exact mechanism of work of HHFNC is not fully explained.The objective of the investigators' research project is to determine the relationship between the amount of airway pressure that can be delivered at specific flow levels of HHFNC. This information will allow the investigators to use HHFNC in a much more informed and safe manner.

DETAILED DESCRIPTION:
Background: Respiratory failure is one of the most common reasons for admission to the Pediatric Critical Care Unit (PCCU). 17% of children admitted to a PCCU require some form of invasive or non-invasive mechanical respiratory support. HHFNC therapy was first introduced in early 2000 and hence is a relatively new mode of respiratory support. One of the proposed mechanisms of action of HHFNC is by providing airway positive pressure hence considered as non-invasive mode of ventilation in pediatrics. However, the actual amount of positive airway pressure that HHFNC provides at increasing flow rates has not been well studied in children.

Objectives: The investigators' objectives are to measure the positive airway pressure delivered with increasing HHFNC flow rates in children, and to evaluate the variables that may influence the delivery of positive airway pressure during HHFNC.

Methods & Design: This is an observational cohort study which will be conducted at McMaster children's hospital, pediatric critical care unit (PCCU). Children under 18 years of age, admitted to PCCU, who require respiratory support by HHFNC, as determined by the caring physician; and informed consent and or assent of substitute decision maker. Those children must have NG tube of size 10 French or smaller inserted at time of HHFNC application. Patients who are on intermittent NGT suction will be excluded. Airway pressure will be measured indirectly using esophageal pressure liquid filled method.

Data Analysis Baseline demographics will be summarized using counts (%) for categorical variables, and mean (standard deviation) or median and interquartile range (IQR) as appropriate for continuous variables. Estimates of the pressure will be reported as mean (95% confidence interval [CI]). Relationship of pressure to delivered flow will be analysed using analysis of variance. Regression methods will be used to determine if the following factors delivered flow per weight of patient, patient size, disease severity, work of breathing and nasal cannula: nares diameter ratio are associated with air pressure

ELIGIBILITY:
Inclusion Criteria:

* Aged less than 18 years, admitted to PCCU with acute respiratory distress.
* HHFNC respiratory support prescribed by the caring physician.
* Requirement for a size 10 French or smaller nasogastric (NG) or orogastric (OG) tube, as prescribed by the caring physician.
* Informed consent, and/- or assent where appropriate.

Exclusion Criteria:

* Continuous or intermittent NG or OG tube suction is required.

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 years, admitted to PCCU, who require respiratory support using HHFNC, as determined by the caring physician; and informed consent of substitute decision maker will be included in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Airway pressure measurement | will be measured at start of HHFNC therapy and with titration of flow rate.
  oesophageal pressure will be measured as a surrogate of airway pressure using Nasogastric tube liquid filled technique.

SECONDARY OUTCOMES:
predictors of positive airway pressure delivery. | will be measured simultaneously with airway pressure
  The secondary outcomes of this study are predictors that may influence the delivery of positive airway pressures during HHFNC, such as the delivered flow per weight of patient, disease severity, work of breathing and nasal cannula: nares diameter ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, FRCP(C), Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada